CLINICAL TRIAL: NCT03246503
Title: BiliCam Clinical Validation Study
Status: Completed | Type: Interventional
Sponsor: BiliCam, LLC (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 52488; R44HD090778 (NIH)
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Results first posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Newborn Jaundice
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Newborns (Experimental): Newborns will be enrolled in the study in 2 different ways. At "Staged Enrollment" sites, newborns will be enrolled when they are < 48 hours old. These newborns will have a study visit when they are 48 - 167 hours old. At the study visit, a BCB will be determined and blood will be drawn for study purposes for a TSB level. At "Simultaneous Enrollment" sites, newborns will be enrolled and have a study visit at the time of a blood draw (+/- 2 hours) for a TSB level that is being obtained for clinical purposes. Newborns will be 0-191 hours old.
  Interventions: Device: BiliCam estimated bilirubin (BCB)

INTERVENTIONS:
Device: BiliCam estimated bilirubin (BCB) — Images will be obtained using the BiliCam app installed on a commercial smartphone and used to calculated a BCB level. The BCB levels will be used for study purposes only and not used for clinical care

SUMMARY:
The goal of this study is to assess the accuracy of BiliCam, a non-invasive technology based on analysis of digital images obtained with an app installed on a commercial smartphone, in estimating total serum bilirubin levels in newborns. BiliCam estimated bilirubin levels will be compared to total serum bilirubin levels in up to 225 newborns.

DETAILED DESCRIPTION:
Jaundice, a yellowing of the skin and eyes caused by a build up of bilirubin in the blood, is a common problem in newborn infants. Measurement of total serum bilirubin (TSB) levels is used for clinical decision making. BiliCam is a non-invasive technology used to estimate TSB levels in newborns. With BiliCam, the user obtains digital images of a small portion of a newborn's skin using the BiliCam app installed on a commercial smartphone in a standardized manner. A color calibration card is placed on the baby's sternum to account for varying light conditions. Data on color levels in the photos are used to estimate a bilirubin level.

For the study, paired BiliCam estimated bilirubin (BCB) and TSB levels will be compared on a racially and ethnically diverse sample of newborns. Recruitment will continue until 225 newborns have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Newborn born at ≥ 35 weeks gestation
* Parent speaks and reads English
* Parent provides written informed consent

Exclusion Criteria:

* previous or ongoing treatment with phototherapy for hyperbilirubinemia
* Medical or other complications that preclude completion of the study

Ages: 0 Hours to 191 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 203 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hopsital, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Newborns
Started | 203
Completed | 150
Not Completed | 53
Not completed — Lost to Follow-up | 23
Not completed — Withdrawal by Subject | 20
Not completed — Physician Decision | 5
Not completed — Received phtototherapy prior to study visit=4, blood specimen not obtained =1 | 5

BASELINE CHARACTERISTICS:
Population: Age was only measured on the 150 participants who completed a study visit
Arm/Group | Newborns
Number analyzed (Participants) | 203
Age, Continuous [Mean (Standard Deviation); unit: hours] — Population: A total of 203 participants were consented. Age was not obtained until the study visit; 150 participants had a study visit
  hours
    number analyzed (Participants) | 150
    (all) | 95.7 (27.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43
  Not Hispanic or Latino | 160
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 61
  White | 80
  More than one race | 39
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 203

OUTCOME MEASURES:

1. Primary Outcome: BCB - TSB Correlation
Description: Pearson correlation coefficient between paired BCB- TSB measurements
Time Frame: Newborns up to 192 hours old
Population: Participants who completed study visit and had valid paired TSB-BCB results. There were 3 participants in whom blood was obtained for TSB levels, but no valid measurement was available (1 grossly hemolyzed sample, 1 specimen lost, and 1 specimen not obtained within 2 hours of the BCB level). There were 3 participants in whom a BCB level could not be obtained by the study device.
Measure: Number; unit: correlation coefficient
Arm/Group | Newborns
Number analyzed (Participants) | 144
correlation coefficient | 0.82
Statistical Analysis 1: Comparison: Newborns; Bootstrapping with 1000 replications was used to estimate 95% confidence intervals; Test type: Other; p < .001, Pearson correlation coefficient — statistical significance of Pearson correlation coefficient; Pearson correlation coefficient = 0.82, 95% CI 2-sided [0.77 to .87] — Bootstrapping with 1000 replications was used to estimate 95% confidence intervals

2. Secondary Outcome: Intercept of Regression Line
Description: The intercept of the regression line of paired BCB TSB values is reported (BCB is the y-axis and TSB is the x-axis).
Time Frame: Newborns up to 192 hours old
Population: Participants with valid paired BCB and TSB values
Measure: Number (95% Confidence Interval); unit: mg/dL
Arm/Group | Newborns
Number analyzed (Participants) | 144
mg/dL | 4.13 [3.35 to 4.91]
Statistical Analysis 1: Comparison: Newborns; Test type: Other — t-statistic from regression analysis; p < .001, Regression, Linear; intercept of regression line = 4.13, 95% CI 2-sided [3.35 to 4.91]

3. Secondary Outcome: Slope of Regression Line
Description: The slope of the regression line of paired BCB TSB values is reported (BCB is the y-axis and TSB is the x-axis).
Time Frame: Newborns up to 192 hours old
Population: Participants with valid paired BCB and TSB values
Measure: Number (95% Confidence Interval); unit: slope
Arm/Group | Newborns
Number analyzed (Participants) | 144
slope | 0.68 [0.60 to 0.76]
Statistical Analysis 1: Comparison: Newborns; Test type: Other — t-statistic from regression analysis; p < .001, Regression, Linear; Slope = 0.68, 95% CI 2-sided [0.60 to 0.76]

ADVERSE EVENTS:
Time Frame: Adverse events related to the study device through study completion, for an average of 30 minutes
Arm/Group | Newborns
All-Cause Mortality (participants affected / at risk) | 0/151
Serious Adverse Events (participants affected / at risk) | 0/151
Other Adverse Events (participants affected / at risk) | 0/151

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT03246503/Prot_SAP_000.pdf